CLINICAL TRIAL: NCT00100009
Title: Multi-Center, Randomized, Phase II/III Clinical Trial to Study the Effects of Preservative-Free Triamcinolone Acetonide as an Adjunct to Photodynamic Therapy in Participants With Neovascular Age-Related Macular Degeneration
Brief Title: Triamcinolone Acetonide Plus Laser Therapy to Treat Age-Related Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050064; 05-EI-0064
Record Dates: First submitted 2004-12-21; First posted 2004-12-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-12-20

CONDITIONS: Macular Degeneration
Keywords: Steroid; Inflammation; Choroidal Neovascularization; Intravitreal Injection; Verteporfin; Age-Related Macular Degeneration; Photodynamic Therapy; Age Related Macular Degeneration; AMD
MeSH Terms: conditions — Macular Degeneration; Inflammation; Choroidal Neovascularization | interventions — Triamcinolone Acetonide

INTERVENTIONS:
Drug: TAC-PF
Drug: Triamcinolone Acetonide

SUMMARY:
This study will test the safety and effectiveness of combining a laser treatment called photodynamic therapy, or PDT, with injections into the eye of the steroid triamcinolone acetonide for treating age-related macular degeneration (AMD). The macula is the part of the retina in the back of the eye that determines central or best vision. AMD can severely impair central vision, affecting a person's ability to read, drive, and carry out daily activities. This vision loss is caused by the formation of abnormal blood vessels behind the retina that leak blood under the macula. PTD stops the growth of these blood vessels and slows the rate of vision loss; however, it has only a temporary effect and does not work in all patients. Furthermore, it may actually cause some swelling and re-growth of blood vessels. Triamcinolone acetonide can help lessen swelling and scarring.

Patients 50 years of age and older with AMD may be eligible for this study. Candidates are screened with a medical history, medical evaluation, and eye examinations (see below). Participants are randomly assigned to one of three treatment groups: 1) PDT plus 1 mg TAC-PF; 2) PDT plus 4 mg TAC-PF; or 3) PDT plus sham injection (a syringe with no needle is pressed against the eye). Treatments are given the day the patient enrolls in the study and then every 3 months for 2 years, as long as the therapy is thought beneficial. Patients who must discontinue TAC-PF injections may still be treated with PDT if medically necessary. In addition to treatment, patients undergo the following tests and procedures:

* Eye examination: Visual acuity and eye pressure are measured, and the lens, retina, pupils and eye movements are examined.
* Fundus photography: Photographs of the back of the eye are taken using a special camera with a bright flash.
* Lens photography: Photographs of the lens are taken to look for development of cataracts.
* Fluorescein angiography: Pictures of the retina are taken to look for abnormal blood vessels. A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. The retina is photographed using a camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible blood vessel abnormality.
* Optical coherence tomography: This test uses light to produce a 2-dimensional cross-sectional picture of the retina. The patient looks into a machine called an optical coherence tomograph at a pattern of flashing and rotating red and green lights, first with one eye and then the other.
* PDT: A needle is placed in an arm vein and a drug called verteporfin (Visudyne® (Registered Trademark)) is infused into the vein over 10 minutes. After 15 minutes, the eye is anesthetized with numbing drops. A special contact lens is then placed on the eye and the laser beam is directed to the eye for 83 seconds.
* TAC-PF or injections (for those in the TAC-PF treatment groups): Numbing and anesthetic drops are placed on the surface of the eye before injection of TAC-PF. Another anesthetic is then applied to the lower part of the eye with a cotton swab. After a few minutes, TAC-PF is injected into the vitreous (jelly-like substance inside the eye). Patients receiving sham injections undergo the identical procedure, except a syringe with no needle is pressed against the eye to seem like a real injection. All patients receive antibiotic drops to put in their eye for 2 days after each treatment. Patients return to the clinic anytime from 2 to 7 days after each treatment for a check of vision, eye pressure, and treatment side effects.

Patients are seen in the clinic for additional checks at 4 weeks and 4 months after the first treatment.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) represents the most common cause of blindness in persons over the age of 50. The major cause of vision loss in this disease is due to the development of choroidal neovascularization. Several clinical trials have shown that eyes with neovascularization portending 4 disc areas or less or all lesions with predominately classic composition (lesions having at least 50% of vessels which can be readily demarcated with fluorescein angiography) can benefit from treatment with photodynamic therapy (verteporfin - PDT). However, this treatment only results in a reduction in the number of participants who suffer moderate and severe vision loss. Few participants demonstrate an improvement in visual acuity.

Histopathologic studies have demonstrated the presence of an inflammatory response in the retina and choroid of participants with choroidal neovascularization as well as in eyes receiving verteporfin - PDT. Therefore, the use of triamcinolone acetonide, which possesses anti-inflammatory as well as anti-angiogenic properties, may be beneficial in participants with neovascular AMD undergoing verteporfin - PDT.

This study will be organized as a controlled, participant masked, randomized, multi-center Phase II/III study that will investigate the efficacy of a preservative - free intravitreal formulation of triamcinolone acetonide (TAC-PF) in AMD participants undergoing verteporfin - PDT. Unlike studies that use steroids containing benzyl alcohol, this study will evaluate preservative-free steroids. Three hundred participants with neovascular AMD, undergoing verteporfin - PDT, will be randomly assigned to receive either a sham intravitreal injection, a 1 mg intravitreal injection of TAC-PF, or a 4 mg intravitreal injection of TAC-PF. Depending on a participant's response, treatments as randomized, may be repeated at 3-month intervals. Participants will complete a maximum of 2 years of follow-up.

The primary efficacy outcome measure is the proportion of participants who experience a moderate vision loss defined as a drop of greater than or equal to 15 letters in best-corrected visual acuity from baseline verteporfin - PDT treatment to month 12. Secondary outcomes will include assessments of the safety of the adjunct therapy; additional vision changes observed between baseline, month 3, month 12, and month 24; lesion changes observed between baseline, month 3, month 12 and month 24; and changes observed in lens opacities between baseline, month 12, and month 24.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for the study, participants must fulfill all of the following criteria:

1. Understand and sign the IRB-approved informed consent document for the study.
2. Age greater than or equal to 50 years.
3. In the study eye, diagnosis of AMD defined by the presence of drusen larger than 63 micro m.
4. In the study eye, participant has had less than three prior pegaptanib sodium (Macugen (Trademark)) injections, without injection-related complications, (such as endophthalmitis, vitreal hemorrhage, or an elevation of IOP greater than or equal to 10 mmHg compared to baseline), the participant's study eye vision is between 20/40 and 20/125, and the last pegaptanib sodium injection occurred greater than 6 weeks prior to randomization.
5. In the study eye, the presence of choroidal neovascularization under the fovea determined by the site Investigator and defined as any one of the following fluorescein angiographic (FA) features:

   1. Early stippled hyperfluorescence of flat retinal pigment epithelium and little or mild leakage in the late frames of the fluorescein (occult).
   2. Irregular elevation of the retinal pigment epithelium that does not exhibit discrete or bright hyperfluorescence in the early transit phase of the angiogram. Stippled hyperfluorescence may be present. Late frames may show persistent fluorescein staining or leakage within a sensory retinal detachment overlying this area (occult).
   3. Late-phase leakage of undetermined source with leakage at the level of the retinal pigment epithelium in the late-phase frames of the angiogram in which the source of the late leakage cannot be determined from earlier-phase frames of the angiogram (occult).
   4. A well-demarcated area of bright hyperfluorescence in the early phase of the angiogram with leakage through the mid- and late-phase frames which obscures the boundaries of the area (classic).
6. For all CNV lesions considered to have occult CNV with no classic CNV, one of the following criteria must be met:

   1. A documented loss of visual acuity (5 or more letters of best-corrected visual acuity if both measurements are made using an ETDRS chart or, a doubling of the visual angle if Snellen acuities are available from either an outside referral center or within the participating center (e.g., 20/80 to 20/160 - a doubling of the visual angle is required because of the measurement variability of Snellen acuities)).

      OR
   2. Documented fluorescein angiographic evidence of a greater than or equal to 10% increase in the lesion greatest linear dimension over the 3 months prior to enrollment.

      OR
   3. Documented blood associated with CNV.
7. The greatest linear dimension of the entire lesion (classic CNV, occult CNV and any features that could obscure the identification of classic or occult CNV) has to be less than or equal to 5400 micro m in greatest linear dimension on the retina as measured by the treating ophthalmologist.
8. Visual acuity of 20/40 - 20/200 (73-34 letter score) as measured on an ETDRS chart.
9. Retinal photographs and angiography of sufficient quality, allowing assessment of the macular area according to standard clinical practice, can be obtained.
10. Women of childbearing potential must not be pregnant or lactating, must have a negative pregnancy test at screening and must be practicing an adequate method of birth control. Acceptable methods of birth control include intrauterine device (IUD); oral, dermal (patch), implanted or injected contraceptives; tubal ligation; and barrier methods with spermicide.
11. Willingness to comply with the protocol.

EXCLUSION CRITERIA:

Participants meeting any of the following criteria will be excluded from the study:

1. Choroidal neovascularization, in the study eye, associated with other ocular diseases such as pathologic myopia, ocular histoplasmosis or posterior uveitis, etc.
2. Presence of geographic atrophy under the fovea in the study eye.
3. Evidence of retinal angiomatous proliferation as suspected by the presence of intraretinal hemorrhage, intraretinal leakage, adjoining serous PED or the presence of a connecting retinal vessel.
4. The presence of a chorio-retinal anastomosis.
5. Decreased vision, in the study eye, due to retinal disease not attributable to CNV, such as nonexudative forms of AMD, geographic atrophy, inherited retinal dystrophy, uveitis or epiretinal membrane. Participants who have any additional ocular diseases that have irreversibly compromised or, during follow-up, could likely compromise the VA of the study eye including amblyopia, anterior ischemic optic neuropathy, clinically significant diabetic macular edema, severe non-proliferative diabetic retinopathy, or proliferative diabetic retinopathy.
6. Decreased vision, in the study eye, due to significant media opacity such as corneal disease or cataract, or opacity precluding photography of the retina; a tear (rip) of the RPE; a vitelliform-like lesion of the outer retina (e.g., as in pattern dystrophies or basal laminar drusen), idiopathic parafoveal telangiectasis, or central serous retinopathy.
7. Presence of fibrosis, hemorrhage, pigment epithelial detachments and other hypofluorescent lesions obscuring greater than 50% of the CNV lesion.
8. History of other antiangiogenic treatment or treatment for CNV (not including photodynamic therapy and pegaptanib sodium injections) in the study eye with transpupillary thermotherapy or other local treatment (such as submacular surgery). Previous laser photocoagulation therapy is acceptable, provided it was not subfoveal.
9. History of photodynamic therapy (PDT) within 1 year of enrollment.
10. Current exam evidence of ocular toxoplasmosis; pseudoexfoliation; external ocular infection, including conjunctivitis; chalazion; significant blepharitis; or aphakia in the study eye (pseudophakic participants are eligible).
11. History of ocular hypertension if intraocular pressure (IOP) is greater than or equal to 25 mm Hg, the participant is on Cosopt with one or more other topical glaucoma medications or is on greater than 2 topical glaucoma medications, not including Cosopt; the most recent visual field, performed within the last 12 months, is abnormal and not attributable to the participant's macular disease; and the optic disc appears glaucomatous.
12. Intraocular surgery (including lens replacement surgery) within 6 weeks prior to randomization.
13. Recent history of (within the last 6 months), or current acute ocular or periocular infection (including any history of ocular herpes zoster or simplex).
14. History of prior treatment with intravitreal corticosteroids.
15. History of peribulbar steroid injection within 6 months prior to randomization.
16. History of oral steroid use at any time during the 30 days prior to randomization.
17. History of untoward complications from corticosteroid therapy, including elevated intraocular pressure in response to topical or periocular corticosteroids that required IOP-lowering treatment.
18. Known hypersensitivity/allergy to verteporfin, porfimer sodium, or other porphyrins, porphyria or other porphyrin sensitivity, or hypersensitivity to sunlight or bright artificial light.
19. Participation in any other clinical study or are receiving, or have received any experimental systemic treatment for AMD (e.g.: retinoic acid, thalidomide) or any other investigational new drug within 12 weeks prior to the start of study treatment.
20. Medical problems that make consistent follow-up over the treatment period unlikely (e.g. stroke, severe MI, end stage malignancy), any contraindications to performing the necessary diagnostic studies (i.e., known allergy to fluorescein dyes, etc.), or in general a poor medical risk because of other systemic diseases or active uncontrolled infections.
21. History of moderate to severe abnormal liver function, unless documented evidence of normal liver enzymes is provided.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-12-09; Study Completion 2006-12-20

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Retina Associates Southwest (RASTA), Tucson, Arizona
  - Doheny Eye Institute, Los Angeles, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Central Florida Retina (CFROL), Orlando, Florida
  - Retina Associates of Florida, Tampa, Florida
  - Midwest Eye Institute, Indianapolis, Indiana
  - Elman Retina Group, P.A. - Baltimore (ERGBM), Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Elman Retina Group, P.A. - Pikesville (ERGPM), Pikesville, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - VitreoRetinal Surgery (VRSMN) Center, Minneapolis, Minnesota
  - Cornell University, New York, New York
  - Duke University Eye Center (DUENC), Durham, North Carolina
  - Dean McGee Eye Institute (DMEIO), Oklahoma City, Oklahoma
  - Casey Eye Institute-Portland, OR (CEIPO), Portland, Oregon
  - Retina Northwest (RNWPO), Portland, Oregon
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Southeastern Retina Associates (SRAKT), Knoxville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Texas Retina Associates, Arlington, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Group of Washington - Fairfax (RGWFF), Fairfax, Virginia
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] BECKER B, MILLS DW. ELEVATED INTRAOCULAR PRESSURE FOLLOWING CORTICOSTEROID EYE DROPS. JAMA. 1963 Sep 14;185:884-6. doi: 10.1001/jama.1963.03060110088027. No abstract available. PMID 14043096